CLINICAL TRIAL: NCT06803134
Title: Effect of Kinetic Control Retraining on Neck Proprioception and Functional Outcome in Patients With Cervical Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ebtesam Wafik Osman Shehab El-Din, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004919
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selected physical therapy program + Kinetic control retraining (Experimental): Participants in this group will be treated by kinetic control retraining for 30 minutes in addition to selected physical therapy program for 30 minutes, 3 sessions per week (day after day), for 8 weeks.
  Interventions: Other: Selected physical therapy program; Other: Kinetic control retraining
- Selected physical therapy program (Active Comparator): Participants in this group will be treated by the same selected physical therapy program for 30 minutes, 3 sessions per week (day after day), for 8 weeks.
  Interventions: Other: Selected physical therapy program

INTERVENTIONS:
Other: Selected physical therapy program — Both groups will receive a selected physical therapy program in the form of trans-cutaneous electrical nerve stimulation (TENS), moist hot pack, posture education, and strengthening exercises for deep neck flexors, for 30 minutes, 3 sessions per week, for 8 weeks.
Other: Kinetic control retraining — Each patient in the experimental group will receive kinetic control retraining for 30 minutes, 3 sessions per week, for 8 weeks. Each session is based on the progression on the motor control rating scale (MCRS) related to kinetic control management frame. For each movement direction, specific control tests will be conducted. The direction and site of the uncontrolled movement will be evaluated using special tests in accordance with the pain history of the patient. The tests will be chosen according to the patient"s symptoms; screening of all patients will be done through at least three tests in each direction according to the patient"s symptoms.
  Arms: Selected physical therapy program + Kinetic control retraining

SUMMARY:
The aim of this study is to investigate the effect of kinetic control retraining on neck proprioception and functional outcome in patients with cervical radiculopathy.

DETAILED DESCRIPTION:
Cervical radiculopathy (CR), which is a normal result of degenerative changes such as cervical disc herniation and bone hyperplasia, is characterized by neck pain and radiating pain from the neck to the shoulder. Neck pain has a major physical, psychological, and socioeconomic impact, as it is the fourth most frequent cause of disability, preceded of low back pain, depression, and arthralgia. In fact, up to 50-70% of the entire population will experience (at least) one episode of neck pain clinically important throughout their life.

Prolonged or recurring stress exposure, pain catastrophism, and fear-avoidance behaviors can trigger variable responses to pain thresholds" intolerance depending on the magnitude of the individual stress response.

Regular physical exercise is a key factor for the prevention of many chronic diseases. Physical exercise (PE) can be used as a primary non-pharmacological clinical tool because it can improve antioxidant capacity, reduce oxidative stress and inflammation and increase energy efficiency. Depending on the volume, the intensity and the frequency of exercise, acute or chronic biochemical and physiological responses are induced. Once movement meets control, they can regain the choices lost in the presence of pain and give people the optimal choice in how they move, these choices are lost with movement impairment. So, the movement value is a central theme in the physical therapy profession and functional concepts which build on movement therapy. These concepts are built on kinetic control approach. This study may add missing information to the existing literature and suggests directions for the effect of kinetic control retraining on neck proprioception and functional outcome in patients with cervical radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Forty Four patients suffering from chronic cervical unilateral radiculopathy (symptomatic duration) (3 months to 1year).
* Their age ranges 40-55 years, from both sexes.
* Body mass index (BMI) of less than 30 Kg/m2
* Cervical spondylosis (at the levels of C5-C6/C6-C7 confirmed by cervical MRI)..

Exclusion Criteria:

* Cervical myelopathy with evidence of pyramidal, posterior column, and or spinothalamic tract lesions.
* Patients with decreased range of motion of cervical spine secondary to congenital anomalies, musculature contracture, or bony block.
* Previous cervical or shoulder surgery or trauma.
* Cervical instability caused by structural problem (e.g. ligament tear or spondylolithesis.
* Psychological problems interfering with the patient understanding of the orders, or patients who did not have direction preference.
* Vertebro-basilar artery insufficiency, diabetic neuropathy.
* Comorbidities that impact physical activity (e.g., cerebrovascular accidents, severe heart disease). - Double crush syndrome and thoracic outlet syndrome.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of cervical proprioception using the cervical range of motion (CROM) device | 8 weeks
  Cervical proprioception will be assessed using the CROM device. Subjects will sit upright in a neutral head position with their trunk and shoulders secured by Velcro straps and will be blindfolded. The CROM unit will be calibrated to zero and secured on the head, with the magnetic yoke positioned on the shoulder. Two tests will be conducted: the Neutral Head Repositioning Test (NHR), where subjects rotate their heads left and return to neutral with accuracy measured in degrees, and the Target Head Repositioning Test (THR), where cervical range of motion will be tested, and subjects will reproduce a memorized target position. Each test will be repeated three times, with average angular displacement error calculated.
Assessment of deep neck flexors (DNFs) strength by craniocervical flexion test (CCFT) using pressure biofeedback unit (PBU) | 8 weeks
  The craniocervical flexion test, a valid and reliable tool for assessing deep neck flexor (DNF) muscle performance, involves positioning the participant in a crook-lying position with a pressure biofeedback unit (PBU) placed under the head. The participant holds the PBU's dial to guide the test, which progresses through five stages based on the pressure exerted at a neutral head position (22, 24, 26, 28, and 30 mmHg). Starting at 20 mmHg, participants perform a slow head nod to incrementally increase the pressure by 2 mmHg, holding each increment for three seconds. Baseline performance is the maximum pressure held correctly for three seconds without substitution, monitored by the tester through palpation of superficial flexors.

SECONDARY OUTCOMES:
Evaluation of neck pain intensity using the Visual Analogue Scale (VAS) | 8 weeks
  The subject will be asked to make a handwritten mark on a 100 mm line (10cm). This line represents a continuum between no pain or discomfort (zero), to the worst pain (10) that the patient could feel. Measurements from the starting point of the scale to the patients' marks will be recorded and interpreted as their pain intensity. The results will be interpreted as: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Evaluation of neck-related functional performance using the Arabic version of Neck Disability Index (NDI) | 8 weeks
  The patient will answer each question by marking the box that best describes their problem, using a six-point scale from 0 (no disability) to 5 (major disability). The total score, out of 50, will be calculated by summing the item scores, with higher scores indicating greater disability. The results will be interpreted as follows: 0-4 = no disability, 5-14 = mild disability, 15-24 = moderate disability, 25-34 = severe disability, and above 34 = complete disability.

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Ahmed Salem, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Horus University, Damietta, Egypt